CLINICAL TRIAL: NCT04203823
Title: Feasibility Study With Personalized Closed Loop (PCL)
Brief Title: Feasibility Studies of Personalized Closed Loop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP326
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single Arm (Cohort) assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Algorithm Testing (Experimental): The main purpose of this cohort is to test the Digital Twin insulin delivery algorithm and the Meal Prediction algorithm
  The study population will be enrolled as 2 separate cohorts to test each algorithms individually
  Interventions: Device: Cloud-based Digital Twin and Meal Prediction algorithms

INTERVENTIONS:
Device: Cloud-based Digital Twin and Meal Prediction algorithms — Test safety and effectiveness of the Digital Twin and Meal Prediction algorithms

SUMMARY:
This is a single arm study comprised of a series of feasibility studies.

DETAILED DESCRIPTION:
Feasibility Study Part 2 (i.e. Feasibility 2): Feasibility 2 is the focus of the current version of the study protocol.

This study will include 2 separate Cohorts of individuals, based on the algorithms being studied:

Cohort A: The main purpose of this cohort is to test the Digital Twin insulin delivery algorithm adaptation

Cohort C: The main purpose of this cohort is to test a meal prediction algorithm

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Subject is age 2-80 years at time of Visit 1. Note: See staged enrollment reference for adult and pediatric subjects in the Study Design section
2. Subject has a clinical diagnosis of type 1 diabetes.

   1. Subjects 7 years of age and older: Diagnosed at least 1 year prior to Visit 1
   2. Subjects 2-6 years of age: Diagnosed at least 3 months prior to Visit 1

   Study-specific inclusion criteria
3. Subject must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units.
4. If subject has a history of hypothyroidism, must have at least 1 documented normal thyroid-stimulating hormone (TSH) on historical labs within 12 months of Visit 1. A subject without a history of hyperthyroidism is not expected to have a TSH test
5. Subjects and their parent(s)/guardian(s) must have Internet access , a computer system that meets the requirements for uploading the study pump and Smartphone that meets study requirements.
6. Subject must have a companion or caregiver available at night for the duration of the study period who resides (or will live) in in the same building (or home). This requirement may be verified by subject report at screening visit.
7. If subject has celiac disease, it has been adequately treated as determined by the investigator.
8. Subjects and their parent(s)/guardian(s) are willing to take one of the following insulins and can financially support the use of either of the 2 insulin preparations throughout the course of the study (i.e. co-payments for insulin with insurance or able to pay full amount)

   * Humalog™* (insulin lispro injection)
   * NovoLog™* (insulin aspart)

Exclusion Criteria:

1. Subject has a history of 1 or more episodes of severe hypoglycemia, which resulted in any the following during the last 1 year prior to Visit 1

   1. Medical assistance (i.e. Paramedics, Emergency Room (ER) or Hospitalization)
   2. Coma
   3. Seizures
2. Subject is unable to tolerate tape adhesive in the area of sensor placement.
3. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
4. Women of child-bearing potential who have a positive pregnancy test at Visit 1 or plan to become pregnant during the course of the study
5. Females who are sexually active and able to conceive will be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
6. Subject has a cardiovascular condition which the Study Investigator determines should exclude the subject, e.g. ventricular rhythm disturbance, hypertrophic cardiomyopathy, recent myocardial infarction in the last year prior to Visit 1.
7. Subject is being treated for hyperthyroidism at time of Visit 1.
8. Subject has a diagnosis of adrenal insufficiency.
9. Subject has had Diabetic Ketoacidosis (DKA) within 1 year prior to Visit 1.
10. Subject has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of visit 1, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
11. Subject is actively participating in an investigational study (e.g., drug or device) wherein he/she has received treatment from an investigational study (drug or device) in the last 2 weeks prior to Visit 1. Please note participation in observational study is acceptable.
12. Subject has been hospitalized or has visited the ER in the 6 months prior to Visit 1 resulting in a primary diagnosis of uncontrolled diabetes.
13. Subject is currently abusing illicit drugs.
14. Subject is currently abusing alcohol.
15. Subject is using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of Visit 1.
16. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
17. Subject has elective surgery planned that requires general anesthesia during the course of the study.
18. Subject diagnosed with current eating disorder such as anorexia or bulimia.
19. Subject has been diagnosed with chronic kidney disease that results in chronic anemia.
20. Subject is on dialysis.
21. Subject has serum creatinine of >2 mg/dL, as confirmed through historical labs within 1 year prior to Visit 1.
22. Subject is a member the research staff involved with the study.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Loma Linda University Medical Center, Loma Linda, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center - Adults, Aurora, Colorado
  - Barbara Davis Center / Pediatric, Aurora, Colorado
  - University of South Florida Diabetes Center, Tampa, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes, Idaho Falls, Idaho
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet International Diabetes Center, Saint Louis Park, Minnesota
  - AM Diabetes and Endocrinology Center, Bartlett, Tennessee
  - Rainier Clinical Research, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: The main purpose of this cohort is to test the Digital Twin insulin delivery algorithm adaptation
  Cloud-based Digital Twin algorithms: Test safety and effectiveness of the Digital Twin algorithms
- Cohort C: The main purpose of this cohort is to test a meal prediction algorithm
  Cloud-based Meal Prediction algorithms: Test safety and effectiveness of the Meal Prediction algorithms
Period: Overall Study
Arm/Group | Cohort A | Cohort C
Started | 54 | 72
Completed | 51 | 65
Not Completed | 3 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Parent/Guardian | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort C | Total
Number analyzed (Participants) | 54 | 72 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (19.2) | 34.8 (19.5) | 35.0 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 28 | 40 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 50 | 62 | 112
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 50 | 69 | 119
  Race: Asian | 1 | 0 | 1
  Race: American Indian or Alaska Native, White | 1 | 0 | 1
  Race: Black or African American | 2 | 1 | 3
  Race: Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 54 | 72 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe Hypoglycemic Event - Cohort A
Description: Number of severe hypoglycemic events occurred in the study in Cohort A
Time Frame: approximately 3.5 months
Measure: Number; unit: events
Arm/Group | Cohort A
Number analyzed (Participants) | 54
events | 0

2. Primary Outcome: Number of Diabetic Ketoacidosis (DKA) Event - Cohort A
Description: Number of Diabetic Ketoacidosis (DKA) event occurred in the study in Cohort A
Time Frame: approximately 3.5 months
Measure: Number; unit: events
Arm/Group | Cohort A
Number analyzed (Participants) | 54
events | 0

3. Primary Outcome: Percentage of Time in Euglycemia - Cohort A
Description: The overall mean percentage of time in Euglycemia (70-180 mg/dL) in Cohort A
Time Frame: approximately 3.5 months
Population: Participants in Cohort A with device data (1 did not have device data)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Cohort A
Number analyzed (Participants) | 53
percentage of time | 70.5 (10.7)

4. Primary Outcome: Number of Severe Hypoglycemic Event - Cohort C
Description: Number of severe hypoglycemic events occurred in the study in Cohort C
Time Frame: approximately 3.5 months
Measure: Number; unit: events
Arm/Group | Cohort C
Number analyzed (Participants) | 72
events | 0

5. Primary Outcome: Number of Diabetic Ketoacidosis (DKA) Event - Cohort C
Description: Number of Diabetic Ketoacidosis (DKA) event occurred in the study in Cohort C
Time Frame: approximately 3.5 months
Measure: Number; unit: events
Arm/Group | Cohort C
Number analyzed (Participants) | 72
events | 0

6. Primary Outcome: Percentage of Time in Euglycemia - Cohort C
Description: The overall mean percentage of time in Euglycemia (70-180 mg/dL) in Cohort C
Time Frame: approximately 3.5 months
Population: Participants in Cohort C with device data (10 did not have device data)
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Cohort C
Number analyzed (Participants) | 62
percentage of time | 77 (8)

ADVERSE EVENTS:
Time Frame: Individual subjects were participating in Feasibility 2 for approximately 3.5 months.
Description: Investigators were instructed to monitor the subjects throughout the course of the study for the occurrence of an adverse event. Adverse events were to be documented in the subject study file and reported to the sponsor on an eCRF. Medtronic study Monitors conducted study site visits and monitored subject source documents to reconcile reported adverse events and for possible detection of additional adverse events.
Arm/Group | Cohort A | Cohort C
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/72
Other Adverse Events (participants affected / at risk) | 14/54 | 22/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=54) | Cohort C (N=72)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2
Immunisation reaction (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Epstein-Barr virus test positive (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT04203823/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04203823/SAP_001.pdf